CLINICAL TRIAL: NCT05452044
Title: A Comparison of Right Ventricular Function in the Apical 4 Chamber and Subcostal 4 Chamber TTE Views in the Perioperative Setting: A Prospective Clinical Study
Brief Title: A Comparison of Right Ventricular Function in the Apical and Subcostal 4 Chamber TTE Views in the Perioperative Setting
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: ID 2020-02841
Record Dates: First submitted 2022-05-18; First posted 2022-07-11 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Assessment of Right Ventricular Function

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators would like to investigate whether angle-independent measurements of the heart's function can be made with the help of new computer programs and modern ultrasound devices. Furthermore, it will be checked whether and to what extent the patient's body position and general anesthesia have an influence on the ultrasound measurements.

DETAILED DESCRIPTION:
Measuring right ventricular function is difficult on account of the ventricles shape, position, and mode of contraction. In transthoracic echocardiography a number of measures are endorsed by current guidelines, including: tricuspid annular plane systolic excursion (TAPSE), tricuspid annular plane velocities (S'), the right ventricular myocardial performance index (MPI), and fractional area change (FAC). Clinically, assessment is usually limited to measuring TAPSE by M-Mode or S' by tissue Doppler imaging, both of which are angle dependent technologies, but unlike the RV MPI or FAC are quick and easy to measure.

In the perioperative period, however, transthoracic echocardiography may be challenging for a number of reasons. First, obtaining usable apical 4-chamber (AP4C) images - the view used to measure TAPSE and S' - may be difficult in ventilated or post-surgical patients; subcostal 4-chamber views (SC4C), however, are generally obtainable. Secondly, gold standard images of the RV function are generally measured in the left lateral decubitus position, rather than supine, as is usually the case perioperative.

Newer technologies - such as speckle-tracking and 3D imaging - may partially overcome these difficulties as these technologies are considered to be relatively angle independent. For example, speckle-tracking can also measure TAPSE and S' and 3D imaging has been shown to correlated very well with MRI, the gold-standard for volume measurements.

This study aims at examining the bias, precision, and reproducibility of speckle-tracking based TAPSE and S' (TAPSESTE and S'STE) measured in the SC4C with measurements of TAPSE by M-Mode and S' TDI (TAPSEM-MODE and S'TDI) in the left lateral decubitus position. Secondly, the investigators will compare measures of RV function made in the supine position to those in the left lateral decubitus position to ascertain the relevance of positioning in the perioperative setting. Patients will have measurements made before and after induction of anaesthesia.

The investigators hypothesize that TAPSE measured by STE in the SC4C with the patient in supine position(TAPSE STE, SC4C, Supine) will be sufficiently similar to TAPSE measured by M-MODE in the AP4C with the patient in the left lateral decubitus position (TAPSE MMODE, AP4C, LLD). A similar hypothesis holds for S' (S' STE, SC4C, Supine and S' TDI, AP4C, LLD).

ELIGIBILITY:
Inclusion Criteria:

* Consenting, adult, in-patients undergoing surgery

Exclusion Criteria:

* Inability to follow the procedures of the study, e.g. due to language problems, vulnerable population, illiterate populations, incompetent/incapacitated adults, -psychological disorders, dementia,
* Previous enrolment into the current study,
* Emergency procedures mandating expeditive patient care,
* Non regular heart rhythm
* Documented valvular heart disease in the RV at least midgrade

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Displacement TAPSE | 25 minutes
  Displacement (TAPSE) measured by:
  TAPSE STE, SC4C, Supine TAPSE MMODE, AP4C, LLD

SECONDARY OUTCOMES:
Velocity (S') | 25 minutes
  TAPSE STE and TAPSEMMODE both in the AP4C, but supine vs. in left lateral decubitus position.
  The effect of frame rate on S'STE measurements

OTHER OUTCOMES:
Reproducibility | 25 minutes
  Correlation of TAPSESTE and S'STE with strain, strain rate, fractional area change (FAC), and right ventricular ejection fraction by 3D.
  Reproducibility of TAPSE and S' measurements by ICC

CONTACTS AND LOCATIONS:
Overall Officials: Eckhard Mauermann, MD, M.Sc, Study Director — University Hospital Basel Department for Anaesthesia
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No
All measurements first are going to be written down on the CRF. After this we are going to enter the data in the system (Redcap®). All written CRF's are then stored in a locked room of the research groups for ten years. After every 10th patient an otherwise uninvolved study nurse will compare the datebase entry in RedCap, the CRF, and the source documents.
  If the findings are insufficient, more frequent checks will occur. Source docs are: premedication documentation, anesthesia record, echo measurement documentation (CRF). These will also be stored in the locked premises of the research group.

REFERENCES:
- See also: Ordinance on Human Research with the Exception of Clinical trials (HRO) — https://www.admin.ch/opc/en/classified-compilation/20121177/index.html
- See also: Human Research Act (HRA) — http://www.admin.ch/opc/en/classified-compilation/20121176/201401010000/810.305.pdf
- See also: Declaration of Helsinki — https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects
- See also: STROBE statement — http://www.jclinepi.com/article/S0895-4356(07)00436-2/pdf